CLINICAL TRIAL: NCT03660475
Title: A Single-Center, Randomized, Double Masked, Placebo Controlled Clinical Study to Assess the Safety and Efficacy of Topical Naltrexone Ophthalmic Solution on the Signs and Symptoms of Dry Eye in Diabetic Subjects
Brief Title: Effect of Topical Naltrexone Ophthalmic Solution on the Signs and Symptoms of Dry Eye in Diabetic Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sassani, Joseph S., MD, MHA (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DDES001/18-110-0002
Record Dates: First submitted 2018-07-18; First posted 2018-09-06 (Actual); Results first posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-10

CONDITIONS: Dry Eye Disease
Keywords: naltrexone; dry eye; diabetic subjects
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Naltrexone (Experimental): Naltrexone Ophthalmic Solution 0.002%
  Interventions: Drug: Naltrexone
- Placebo (Placebo Comparator): Placebo Ophthalmic Solution
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Naltrexone — naltrexone formulated as ophthalmic solution
  Arms: Naltrexone
Drug: Placebos — Placebo ophthalmic solution
  Arms: Placebo

SUMMARY:
The objective of this exploratory study is to determine the safety and efficacy of 0.002% Naltrexone Ophthalmic Solution, compared to placebo for the treatment of the signs and symptoms of dry eye in diabetic subjects.

DETAILED DESCRIPTION:
This is a Phase 2, single-center, double-masked, randomized, placebo-controlled study to compare the safety and efficacy of Naltrexone Ophthalmic Solution, 0.002% to placebo for the treatment of the signs and symptoms of dry eye in diabetic subjects. Subjects eligible to be randomized will receive one of the following treatments to be administered bilaterally BID for 29 days (from Visit 2 to Visit 5): Naltrexone Ophthalmic Solution, 0.002% or Placebo Ophthalmic Solution (Vehicle). During a 10-day study run-in period (for the purpose of subject selection) prior to randomization, all subjects will receive Placebo Ophthalmic Solution (Vehicle) bilaterally BID. Participants who terminate early during the application period will be asked to complete safety assessments (if the participants agree) prior to study exit. Participants who are terminated early from the study will not be replaced.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent;
* Have a diagnosis of type 1 or type 2 diabetes mellitus prior to Visit 1;
* Have a reported history of dry eye for at least 6 months prior to Visit 1;
* Have a history of use or desire to use eye drops for dry eye symptoms within 6 months of Visit 1;
* Have a corneal fluorescein staining score of ≥ 2 in any region (inferior, superior, or central regions) in at least one eye at Visits 1 and 2 (must be the same eye at Visits 1 and 2);
* Have at least one of the following at Visits 1 and 2:

  1. A total lissamine green conjunctival score of ≥ 2 in at least one eye, based on the sum of the temporal and nasal regions at Visits 1 and 2 (must be the same eye at Visits 1 and 2);
  2. Report an OSDI score ≥ 20 at Visits 1 and 2.

Exclusion Criteria:

* Have any clinically significant slit lamp findings at Visit 1 that may include active blepharitis, meibomian gland dysfunction (MGD), lid margin inflammation or active ocular allergies that require therapeutic treatment, and/or in the opinion of the investigator may interfere with study parameters;
* Be diagnosed with an ongoing ocular infection (bacterial, viral, or fungal), or active ocular inflammation at Visit 1;
* Have concurrent neurotrophic keratopathy from a source other than diabetes (h/o HSV keratitis, h/o HZO with ocular manifestations, or CN VII palsy or other condition resulting in lagophthalmos);
* Have active diabetic foot ulcers;
* Have a corneal sensitivity score ≤ 1.5 cm as measured by Cochet-Bonnet at Visit 1;
* Report an OSDI score > 75 at Visits 1 and 2;
* Have worn contact lenses within 21 days of Visit 1 or anticipate using contact lenses during the study (no contact lens wear during study);
* Have used any eye drops within 2 hours of Visit 1;
* Have previously had laser-assisted in situ keratomileusis (LASIK) surgery within the last 24 months;
* Have used cyclosporine 0.05% or lifitigrast 5.0% ophthalmic solution within 45 days of Visit 1;
* Have any planned ocular and/or lid surgeries over the study period or any ocular surgery within the last 12 months;
* Be using or anticipate using temporary punctal plugs during the study that have not been stable within 30 days of Visit 1;
* Be currently taking any topical ophthalmic prescription (including medications for glaucoma) or over-the-counter (OTC) solutions, artificial tears, gels or scrubs, and cannot discontinue these medications for the duration of the trial (excluding medications allowed for the conduct of the study);
* Have corrected visual acuity greater than or equal to logMAR +0.7 as assessed by Early Treatment of Diabetic Retinopathy Study (ETDRS) scale in either eye at Visit 1;
* Have concurrent autoimmune disease causing dry eye (e.g., rheumatoid arthritis, Sjogren's, GVHD, Steven's Johnson, Grave's);
* Have Fuchs endothelial dystrophy;
* Have recurrent corneal erosion syndrome or anterior basement membrane dystrophy;
* Be a woman who is pregnant, nursing, or planning a pregnancy;
* Be unwilling to submit a urine pregnancy test at Visit 1 and Visit 5 (or early termination visit) if of childbearing potential. Non-childbearing potential is defined as a woman who is permanently sterilized (i.e., has had a hysterectomy or bilateral tubal ligation), or is post-menopausal (without menses for 12 consecutive months);
* Be a woman of childbearing potential who is not using an acceptable means of birth control; acceptable methods of contraception include: hormonal - oral, implantable, injectable, or transdermal contraceptives; mechanical - spermicide in conjunction with a barrier such as a diaphragm or condom; IUD; or surgical sterilization of partner. For non-sexually active females, abstinence may be regarded as an adequate method of birth control; however, if the subject becomes sexually active during the study, they must agree to use adequate birth control as defined above for the remainder of the study;
* Have a known allergy and/or sensitivity to the test article or its components;
* Have a condition or be in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study;
* Be currently enrolled in an investigational drug or device study or have used an investigational drug or device within 30 days of Visit 1;
* Be currently using any medication known to cause ocular drying that is not used on a stable dosing regimen for at least 30 days prior to Visit 1;
* Be unable or unwilling to follow instructions, including participation in all study assessments and visits.
* Be currently using a systemic opioid antagonist (e.g., Naltrexone or Naloxone) or have used a systemic opioid antagonist in the previous 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene B McLaurin, M.D., Principal Investigator — Total Eye Care
Locations (1):
- Total Eye Care, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty subjects (30 subjects per treatment arm) were planned. For this number, it was anticipated that 120 subjects would be screened. A total of 87 subjects were screened to enroll 60 subjects who were analyzed for efficacy and safety.
Period: Overall Study
Arm/Group | Naltrexone | Placebo
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naltrexone | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.64 (7.86) | 62.64 (10.97) | 64.14 (9.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 13 | 12 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 21 | 41
  White | 10 | 9 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Total Ocular Surface Disease Index
Description: The OSDI is a 12-item questionnaire designed to provide a rapid assessment of the symptoms of ocular irritation consistent with dry eye disease and their impact on vision-related functioning. It is a scale of 0-4 for each of the 12 questions. A minimum value would be "0" and a maximum value would be "48". The higher the value the worse the outcome.
Time Frame: Day 29
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 30 | 30
score on a scale | 21.17 (17.72) | 21.36 (17.16)
Statistical Analysis 1: Comparison: Naltrexone vs Placebo; Test type: Superiority; p = 0.967, t-test, 2 sided

2. Secondary Outcome: Lissamine Green Staining
Description: Lissamine green staining; regions: inferior, superior, central, corneal sum, temporal, nasal, conjunctival sum, total eye will be measured using an ocular discomfort score on a scale of 0 (no staining) to 4 (confluent staining). The total eye score is presented. A minimum score would be "0" and a maximal score would be "8". The higher the value the worse the outcome.
Time Frame: Day 29
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 30 | 30
score on a scale | 2.65 (1.10) | 2.59 (1.25)
Statistical Analysis 1: Comparison: Naltrexone vs Placebo; Test type: Superiority; p = 0.836, t-test, 2 sided

3. Secondary Outcome: Tear Film Break-up Time
Description: Tear film break-up time is the time taken for the first dry spot to appear on the cornea after a complete blink.
Time Frame: Day 29
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 30 | 30
seconds | 2.76 (0.98) | 3.48 (2.49)
Statistical Analysis 1: Comparison: Naltrexone vs Placebo; Test type: Superiority; p = 0.166, t-test, 2 sided

4. Secondary Outcome: Conjunctival Redness
Description: Conjunctival redness will be assessed and conjunctival pain will be assessed using a visual analog scale ranging from "0" (none: normal without vasodilation) to "5" (severe: broad ciliary and prominent, horizontal conjunctival vasodilation). A minimal score would be "0" and a maximal score would be "10". The higher the value the worse the outcome .
Time Frame: Day 29
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 30 | 30
score on a scale | 1.0 (0.41) | 1.0 (0.45)
Statistical Analysis 1: Comparison: Naltrexone vs Placebo; Test type: Superiority; p = 0.638, t-test, 2 sided

5. Secondary Outcome: Schirmer's Test
Description: Schirmer's Test (without anesthesia) ) involves placing a Schirmer test strip in the lower temporal lid margin of each eye such that the strip fits tightly. Subjects will be instructed to close their eyes. After 5 minutes have elapsed, the Schirmer strip will be removed. The length of the moistened area will be recorded (mm) for each eye. A normal reading is ≥10 mm wetting of the paper after 5 minutes. Tear deficiency is <5 mm wetting of the paper after 5 minutes.
Time Frame: Day 29
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 30 | 30
mm | 8.97 (8.00) | 12.48 (9.20)
Statistical Analysis 1: Comparison: Naltrexone vs Placebo; Test type: Superiority; p = 0.122, t-test, 2 sided

6. Secondary Outcome: Cochet-Bonnet Corneal Sensitivity Test
Description: After extending the Cochet-Bonnet corneal sensitivity device (containing a thin, retractable, nylon monofilament) up to 6 cm in length and pressing against the cornea, the monofilament is slowly retracted incrementally in 0.5 cm steps until the patient can feel its contact and the length is recorded. The greater the length indicates increased sensation and the shorter the length indicates decreased sensation.
Time Frame: Day 29
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 30 | 30
cm | 59.78 (0.95) | 59.37 (1.44)
Statistical Analysis 1: Comparison: Naltrexone vs Placebo; Test type: Superiority; p = 0.200, t-test, 2 sided

7. Secondary Outcome: Tear Osmolarity
Description: Normal tear osmolarity is defined as < 300 mOsm/L in both eyes and an inter-eye difference of < 8 mOsm/L. Values greater than 300 mOsm/L are suggestive of dry eye.
Time Frame: Day 29
Measure: Mean (Standard Deviation); unit: mOsm/L
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 30 | 30
mOsm/L | 304.31 (14.11) | 310.66 (12.16)
Statistical Analysis 1: Comparison: Naltrexone vs Placebo; Test type: Superiority; p = 0.085, t-test, 2 sided

8. Secondary Outcome: Matrix Metalloprotienase-9 (MMP-9) is a Marker of Inflammation.
Description: Levels of MMP-9 will be measured in each eye using InflammaDry at Visit 5. The test will be recorded as either positive or negative. Dry eye patients generally exhibit positive levels of MMP-9., so the number of subjects testing positive for MMP-9 at Day 29 will be recorded.
Time Frame: Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 30 | 30
Participants | 3 | 3

9. Secondary Outcome: Ocular Discomfort (Scale 1)
Description: Ocular discomfort scores will be subjectively graded by the subjects according to the following scale, rating each eye separately on a scale from 0-4. A score of "0" represents no discomfort and a score of "4" represents constant discomfort. A minimum score would be "0" and a maximum score would be "8". The higher the value the worse the outcome.
Time Frame: Day 29
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 30 | 30
score on a scale | 1.03 (1.10) | 1.07 (1.13)
Statistical Analysis 1: Comparison: Naltrexone vs Placebo; Test type: Superiority; p = 0.903, t-test, 2 sided

10. Secondary Outcome: Ocular Discomfort (Scale 2)
Description: Subjects will rate the severity of each of the following symptoms, with regard to how both their eyes feel: overall ocular discomfort, burning, dryness, grittiness and stinging according to the following 6-point (0 to 5) scale where 0 = none and 5 = worst. A minimum score would be "0" and a maximum score would be "10". The higher the value the worse the outcome.
Time Frame: Day 29
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 30 | 30
score on a scale | 1.40 (1.25) | 1.45 (1.57)
Statistical Analysis 1: Comparison: Naltrexone vs Placebo; Test type: Superiority; p = 0.898, t-test, 2 sided

11. Secondary Outcome: Visual Analog Scale for Pain
Description: Standard scale assessing a patient's level of pain on a scale of 0-100. The subject will be asked to rate each ocular symptom due to ocular dryness by placing a vertical mark on the horizontal line to indicate the level of discomfort. 0% corresponds to "no discomfort" and 100% corresponds to "maximal discomfort". The following parameters will be assessed: burning/stinging, itching, foreign body sensation, blurred vision, eye dryness, photophobia, and pain, with a total score for each eye reported. A minimal score would be "0" and a maximum score would be "200". The higher the value the worse the outcome.
Time Frame: Day 29
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 30 | 30
score on a scale | 16.27 (22.82) | 25.07 (31.32)
Statistical Analysis 1: Comparison: Naltrexone vs Placebo; Test type: Superiority; p = 0.221, t-test, 2 sided

12. Secondary Outcome: Fluorescein Staining
Description: The following regions of each eye will be assessed for fluorescein staining: inferior, superior, central, corneal sum, temporal, nasal, conjunctival sum, and a total eye score recorded. A score of "0" represents no staining and a score of "4" represents confluent staining. A minimum score would be "0" and a maximum score would be "8". A higher values represent a worse outcome.
Time Frame: Day 29
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 30 | 30
score on a scale | 7.70 (2.53) | 7.14 (3.23)
Statistical Analysis 1: Comparison: Naltrexone vs Placebo; Test type: Superiority; p = 0.459, t-test, 2 sided

13. Secondary Outcome: Visual Acuity Measured by Assessing Average Change in LogMAR Units for Both Eyes at Day 29. LogMAR Units Range From 0-1.0, With the Higher the Number Indicating a Worsening in Vision.
Description: Mean change in visual acuity (LogMAR units 0-1.0) for both eyes at Day 29 was determined for each treatment arm and considered a measure of safety.
Time Frame: Day 29
Population: Mean change in visual acuity for both eyes measured by LogMAR units (0-1.0)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 30 | 30
units on a scale | 0.08 (0.11) | 0.07 (0.13)

14. Other Pre Specified Outcome: Number of Participants With Treatment-related Adverse Events
Description: An adverse event is defined as any untoward medical occurrence associated with the use of the investigational agent (or placebo) regardless of whether or not it is considered related to the investigational drug (or placebo).
Time Frame: Adverse events will be collected from first dose of study drug to 30 days after treatment discontinuation (Day 29 + 4 weeks).
Measure: Count of Participants; unit: Participants
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 30 | 30
Participants | 0 | 1

15. Other Pre Specified Outcome: Slit-lamp Biomicroscopy
Description: The binocular slit-lamp examination provides a stereoscopic magnified view of the eye structures in detail, enabling anatomical diagnoses to be made of the cornea, conjunctiva, anterior chamber, iris, lens and lid for both eyes. The number of subjects in each treatment arm that have changes in the cornea, conjunctiva, anterior chamber, iris, lens and lid for both eyes at Day 29 will be reported.
Time Frame: Day 29
Measure: Number; unit: participants
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 30 | 30
participants | 0 | 0

16. Other Pre Specified Outcome: Intraocular Pressure
Description: Intraocular pressure is the fluid pressure inside the eye.
Time Frame: Day 29
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 30 | 30
mmHg | 14.95 (3.30) | 14.65 (2.90)

17. Other Pre Specified Outcome: Dilated Fundoscopy
Description: Dilated fundus examination is a diagnostic procedure that employs the use of mydriatic eye drops to dilate the pupil in order to obtain a better view of the fundus of the eye. The number of subjects that demonstrate clinically significant abnormalities in the vitreous, choroid, macula, and optic nerve at Day 29 in either treatment arm will be reported.
Time Frame: Day 29
Measure: Number; unit: participants
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 30 | 30
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Through Day 29 + four week follow-up period
Description: Deaths and adverse events were not reported on during the Run-In Period
Arm/Group | Naltrexone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 1/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Naltrexone (N=30) | Placebo (N=30)
Swelling of upper lip (Skin and subcutaneous tissue disorders) | 0 | 1
Increase in A1C (Metabolism and nutrition disorders) | 0 | 1
Rotator cuff pain (Musculoskeletal and connective tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Please note that no specific primary endpoint was identified in the protocol. The study was exploratory in nature looking at both efficacy and safety parameters to help inform future studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/75/NCT03660475/Prot_SAP_001.pdf